CLINICAL TRIAL: NCT04610255
Title: Effects of Dynamic Myofascial Release in Patients With Non-specific Neck Pain.
Brief Title: Dynamic Myofascial Release in Patients With Non-specific Neck Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00678 Haseeb Shah
Record Dates: First submitted 2020-10-09; First posted 2020-10-30 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Neck Pain
Keywords: Neck Pain; Myofascial Release; Dynamic Myofascial Release
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional physical therapy (Active Comparator): Cervical isometrics and Muscle Stretching
  Interventions: Other: Assigned Interventions
- Dynamic myofascial release (Experimental): Experimental group was given Dynamic myofascial release along with the cervical isometrics and muscle stretching
  Interventions: Other: Dynamic myofascial release

INTERVENTIONS:
Other: Assigned Interventions — * Hot pack for 10 minutes
  * TENS for 10 minutes
  * Trigger point release if any found.
  * Myofascial release
  * Home plan for stretching exercises will be prescribed to the patient. Receive two weeks intervention plan, three sessions per week.
  Arms: Traditional physical therapy
Other: Dynamic myofascial release — DMFR involves a manual application of low amplitude, long duration stretch to the fascia and muscle. Participants were instructed to relax as much as possible, and the therapist proceeded to smoothly move the joints in a diagonal or horizontal direction at a slow rate within the ROM. The therapist repeatedly pushed, pulled, or shook the joint area about three to five times for about 3 seconds with slight motion at the end of ROM.
  Conventional therapy will includes
  * Hot pack for 10 minutes
  * TENS for 10 minutes
  * Trigger point release if any found.
  * Myofascial release
  * Home plan for stretching exercises will be prescribed to the patient. Receive two weeks intervention plan, three sessions per week.
  Arms: Dynamic myofascial release

SUMMARY:
Dynamic myofascial release is similar to joint mobilization (active physiological movements) to increase ROM with the myofascial release for fascia release. It differs from myofascial release in a way that it is a dynamic approach in which the patient is actively involved. In 2019 study was conducted on the effects of Dynamic myofascial release showing significant increase in all trunk ROMs and functional reach test in patients with chronic non-specific low back pain.

To summarize, this study will going to see the effectiveness of dynamic myofascial release by addressing both fascia and active physiological movements and see the response of patient's pain level, cervical ROM, improvement in the ability to manage in activities of daily life. Furthermore this study helps to find out its effectiveness and its clinical importance in treating patients with neck pain, considering its significance of engaging multiple structures.

DETAILED DESCRIPTION:
Neck pain is one of the most common and painful musculoskeletal conditions. For the majority of the neck disorders there is an absence of an identifiable underlying disease or abnormal anatomical structure. As a consequence they are classified as 'non-specific'. The natural course of nonspecific neck pain remains unclear. While it is often self-limiting within a few weeks of onset, it can severely limit daily functioning, induce substantial medical consumption and result in prolonged sick leave and disability. As a consequence it places a heavy burden on individuals, employers and health care services." Non-specific neck pain, also referred to as mechanical neck pain, is diagnosed as cervical pain with or without radiation without a known pathological basis as the underlying cause of the complaints.Overall analysis revealed evidence that middle age and then adults, female gender, high job demands, low social or work support, being an ex-smoker, a history of low back disorders and a history of neck disorders predicts the future onset of neck pain.

In recent years, several studies have emerged about myofascial pain syndrome among patients suffering from neck pain. Myofascial pain syndrome is the presentation of sensory, motor, and autonomic symptoms caused by Myofascial trigger points . In 2014 study concluded that the most prevalent active myofascial trigger points in the trapezius muscles were identified in 93.75% of the subjects, in the levator scapulae in 82.14%, and in the multifidi in 77.68% of the subjects. Myofascial trigger points in the splenius cervicis reached a prevalence of 62.5% .

Myofascial release is a widely employed manual therapy treatment that involves specifically guided low load, long duration mechanical forces to manipulate the myofascial complex, intended to restore optimal length, decrease pain, and improve function. Myofascial release when used in conjunction with conventional treatment is said to be effective to provide immediate relief of pain and tissue tenderness.

Myofascial release generally involves slow, sustained pressure applied to restricted fascial layers either directly (direct MFR technique) or indirectly (indirect MFR technique). Direct Myofascial release technique is thought to work directly over the restricted fascia: practitioners use knuckles or elbow or other tools to slowly sink into the fascia, and the pressure applied is a few kilograms of force to contact the restricted fascia, apply tension, or stretch the fascia. Indirect Myofascial release involves a gentle stretch guided along the path of least resistance until free movement is achieved.

In 2018 study concluded in a study to see the effects of Myofascial release in patients with neck pain that both Myofascial release and Physical therapy multimodal programs provide improvement of pain in patients with neck pain. However, Myofascial release could be better than a Physical therapy multimodal program that includes Ultrasound , TENS, and massage. Overall, the improvement of pressure pain threshold provided by MFR was 20% greater than that provided by a Physical therapy multimodal program. In 2017 study found significant improvement in both pain and disability among patients with low back pain in response to myofascial release applied to the lumbar region. In 2018 study performed Myofascial release on thoracic spine and demonstrated that Myofascial release can be effective in increasing both local and distal Range of motion.

ELIGIBILITY:
Inclusion Criteria:

* Participants had a complaint of non-specific pain in the neck with duration of at least 3 weeks.
* The area of neck pain was defined to the cervical Region, with or without radiating to head or arms.
* Patients with tight upper trapezius or levator scapulae or both with or without the presence of myofascial trigger points.

Exclusion Criteria:

* NP due to traumatism, fractures, or whiplash;
* Neoplasia, severe osteoporosis, infectious, or inflammatory processes.
* Ppatient's with pacemakers, congenital anomalies, previous neck surgery, or pregnancy.
* Patients who had received MRT in the previous month.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
Numeric pain rating scale | 2 weeks
  The NPRS can be administered verbally or graphically for self-completion. The respondent is asked to indicate the numeric value on the segmented scale that best describes their pain intensity. High test-retest reliability has been observed (r = 0.96 and 0.95, respectively with minimum score 0 to maximum 10

SECONDARY OUTCOMES:
Inclinometer | 2 weeks
  The instrument has an inclination needle, affected by gravity that is used to measure ranges of cervical spine, with ICCs ranging from .89 to .94
Neck Disability Index | 2 weeks
  The Neck Disability Index (NDI) is a 10-item questionnaire that measures a patient's self-reported neck pain related disability. It has been shown to have high "test-retest" reliability. The NDI has also been shown to be valid when comparing it to other pain and disability measures. Each of the 10 items is scored from 0 - 5. The maximum score is therefore 50

CONTACTS AND LOCATIONS:
Overall Officials: Shafaq Shahid, MSPT(OMPT), Principal Investigator — Riphah International University
Locations (1):
- Maroof International Hospital, Islamabad, Fedral,Pakistan, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cerezo-Tellez E, Torres-Lacomba M, Mayoral-Del Moral O, Sanchez-Sanchez B, Dommerholt J, Gutierrez-Ortega C. Prevalence of Myofascial Pain Syndrome in Chronic Non-Specific Neck Pain: A Population-Based Cross-Sectional Descriptive Study. Pain Med. 2016 Dec;17(12):2369-2377. doi: 10.1093/pm/pnw114. Epub 2016 Jun 20. PMID 28025371
- [Background] McLean SM, May S, Klaber-Moffett J, Sharp DM, Gardiner E. Risk factors for the onset of non-specific neck pain: a systematic review. J Epidemiol Community Health. 2010 Jul;64(7):565-72. doi: 10.1136/jech.2009.090720. Epub 2010 May 12. PMID 20466711
- [Background] Ajimsha MS, Al-Mudahka NR, Al-Madzhar JA. Effectiveness of myofascial release: systematic review of randomized controlled trials. J Bodyw Mov Ther. 2015 Jan;19(1):102-12. doi: 10.1016/j.jbmt.2014.06.001. Epub 2014 Jun 13. PMID 25603749
- [Background] Rodriguez-Huguet M, Lomas-Vega R. Response to the Letter to the Editor on "Effects of Myofascial Release on Pressure Pain Thresholds in Patients With Neck Pain: A Single-Blind Randomized Controlled Trial". Am J Phys Med Rehabil. 2019 Jan;98(1):e4-e5. doi: 10.1097/PHM.0000000000000986. No abstract available. PMID 29912003
- [Background] Arguisuelas MD, Lison JF, Sanchez-Zuriaga D, Martinez-Hurtado I, Domenech-Fernandez J. Effects of Myofascial Release in Nonspecific Chronic Low Back Pain: A Randomized Clinical Trial. Spine (Phila Pa 1976). 2017 May 1;42(9):627-634. doi: 10.1097/BRS.0000000000001897. PMID 28441294
- [Background] Cathcart E, McSweeney T, Johnston R, Young H, Edwards DJ. Immediate biomechanical, systemic, and interoceptive effects of myofascial release on the thoracic spine: A randomised controlled trial. J Bodyw Mov Ther. 2019 Jan;23(1):74-81. doi: 10.1016/j.jbmt.2018.10.006. Epub 2018 Oct 24. PMID 30691766
- [Background] Ferraz MB, Quaresma MR, Aquino LR, Atra E, Tugwell P, Goldsmith CH. Reliability of pain scales in the assessment of literate and illiterate patients with rheumatoid arthritis. J Rheumatol. 1990 Aug;17(8):1022-4. PMID 2213777
- [Background] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748